CLINICAL TRIAL: NCT06309368
Title: To Close or Not to Close: Surgical Site Infection Rates in Ostomy Primary Closure With 0.1% Betaine/Polyhexanide Wound Irrigation Compared to Conventional Ostomy Closure by Secondary Intention
Brief Title: Ostomy Primary Closure With 0.1% Betaine/Polyhexanide Wound Irrigation Compared to Pursestring Closure
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Ovunc Bardakcioglu, Chief of Colorectal Surgery, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003875
Record Dates: First submitted 2024-02-22; First posted 2024-03-13 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Surgical Site Infection; Wound Surgical; Colorectal Disorders
Keywords: Ostomy; Surgical Site Infection; Primary Closure; Secondary Closure
MeSH Terms: conditions — Surgical Wound Infection; Surgical Wound

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two treatment groups.
Masking Description: No masking. This is a non-blinded randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary Closure with 0.1% Betaine/0.1% Polyhexanide Wound Irrigation (Active Comparator): The ostomy wound will be irrigated with 0.1% Betaine/0.1% Polyhexanide wound irrigation, then closed completely with sutures.
  Interventions: Drug: Primary Ostomy Closure with 0.1% Betaine/0.1% Polyhexanide Wound Irrigation
- Secondary Closure with Pursestring (Active Comparator): The ostomy wound will be partially closed using the Pursestring method.
  Interventions: Procedure: Pursestring Closure

INTERVENTIONS:
Drug: Primary Ostomy Closure with 0.1% Betaine/0.1% Polyhexanide Wound Irrigation — An elliptical transverse incision will be made extending 1-2 cm lateral and medial to the mucocutaneous junction. The mobilization, anastomosis and fascial closure will be performed as in the pursestring closure group. The incision will then be irrigated using direct stream into the wound with 350cc of Prontosan. After one minute the wound will be suctioned dry. The subcutaneous fat will be mobilized and approximated with interrupted 2-0 Vicryl. The skin will be approximated with deep dermal 3-0 Vicryl and a running subcuticular 4-0 Monocryl suture and Dermabond will be applied.
  Other Names: Prontosan
  Arms: Primary Closure with 0.1% Betaine/0.1% Polyhexanide Wound Irrigation
Procedure: Pursestring Closure — A circular incision will be made at the mucocutaneous junction of the ileostomy. After complete mobilization of the ileal limbs off the fascia and a stapled side to side functional end to end anastomosis, the fascia including the external and posterior rectus sheath will be closed with two running #0 PDS (Polydioxanone) suture. The wound will then be irrigated with saline and partially closed in the subcuticular plane with a 2-0 Monocryl suture in a pursestring fashion and packed in the middle with plain packing.
  Arms: Secondary Closure with Pursestring

SUMMARY:
The goal of this clinical trial is to compare two types of closure in patients with ostomies that are ready for closure. The main questions it aims to answer are:

1. Surgical site infection rates
2. Patient quality of life
3. Time to wound healing

Participants will undergo either complete ostomy wound closure after washing out the wound with Prontosan, or their ostomy wound will be closed using the Pursestring method, where the wound will be left partially open and allowed to heal from the inside out. Researchers will compare these two groups' outcomes (questions to be answered) as listed above.

DETAILED DESCRIPTION:
Surgical site infection (SSI) is a common yet potentially serious and devastating complication in colorectal surgery, with rates of up to 25%, many of which are preventable. In stoma closure, SSI rates have been reported as up to 40% with conventional closure techniques. SSI adds more burden to the patient, requiring additional therapy, such as antibiotics, wound drainage, and even wound debridement. This results in longer hospital length of stay and can ultimately negatively impact a patient's quality of life. Additionally, allowing a wound to heal by secondary intention has been demonstrated to have worse cosmetic outcomes compared to primary closure, which may also impact quality of life (QoL) for patients. The investigators aim to investigate the outcomes (including SSI rates and QoL) of patients who underwent two different standards of care in ostomy closure: primary skin closure after usage of Prontosan, a 0.1% betaine and 0.1 % polyhexamethylene biguanide antimicrobial solution, and secondary intention healing after Pursestring closure. Comparing these two closure methods, may yield further insight into better treatment options for wound closures in colorectal surgery patients.

Patients will be recruited in the UNLV Colorectal Clinic at their appointments, and surgeries will be done at University Medical Center. Patient recruitment and informed consent will be performed by the co-investigators. The sample size is calculated for a non-inferiority trial with a 2.5% level of significance, 90% power of test and an expected SSI rate of 3% for the purse-string closure group and 25.9% for the primary wound closure without 0.1% betaine/0.1% polyhexanide). The sample size needed is 42 patients in each study arm with an assumed 20% attrition rate. Data will be analyzed by the statistician.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years or older with an diverting loop ileostomy reversal indication will be enrolled
* Signed consent

Exclusion Criteria:

* Under 18 years old, unable to provide consent, has a parastomal hernia requiring mesh repair, or has an end ileostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection Rates | Evaluate surgical site for any signs of infection up to 30 days post-operatively.
  Evaluate surgical site infection rates between the two treatment arms

SECONDARY OUTCOMES:
Acceptability of wound or scar healing by patient | Up to one year post-operatively.
  Evaluation of patient's perception of their ostomy wound or scar appearance using the Visual Analog Scale. The minimum value is 0, maximum value is 10, with the higher score meaning a worse outcome.
Amount of percepted wound care needed by patient | Up to 4 weeks after compete wound closure.
  Evaluation of patient's perception of the amount of wound care needed during the healing of their ostomy wound using the Visual Analog Scale. The minimum value is "no wound care needed" and maximum value is "maximum amount of wound care needed", with "maximum amount of wound care needed" being the worst outcome.
Acceptability of wound and scar healing by patient | At 4 weeks post complete wound closure and at one year post-operatively.
  Evaluation of patient's perception of their ostomy wound and scar appearance using the Patient and Observer Scar Assessment Scale - Observer scale. The minimum value is 1 and maximum value is 10, with the higher score meaning a worse outcome.
Wound healing | Until complete wound closure (estimated up to 4-6 weeks post-operation).
  Time to wound-healing
Acceptability of wound and scar healing by patient | Up to one year post-operatively
  Evaluation of patient's satisfaction of their ostomy wound and scar appearance using the Likert Scale. The minimum value is "very dissatisfied" and maximum value is "very satisfied", with "very satisfied being the best outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ovunc Bardakcioglu, MD, Principal Investigator — Kirk Kerkorian School of Medicine at UNLV
Locations (1):
- University Medical Center, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Cooper DM, Bojke C, Ghosh P. Cost-Effectiveness of PHMB & betaine wound bed preparation compared with standard care in venous leg ulcers: A cost-utility analysis in the United Kingdom. J Tissue Viability. 2023 May;32(2):262-269. doi: 10.1016/j.jtv.2023.03.001. Epub 2023 Mar 16. PMID 36990897
- [Background] Valenzuela AR, Perucho NS. [The effectiveness of a 0.1% polyhexanide gel]. Rev Enferm. 2008 Apr;31(4):7-12. Spanish. PMID 18564781
- [Background] Siddiqi A, Abdo ZE, Springer BD, Chen AF. Pursuit of the ideal antiseptic irrigation solution in the management of periprosthetic joint infections. J Bone Jt Infect. 2021 May 26;6(6):189-198. doi: 10.5194/jbji-6-189-2021. eCollection 2021. PMID 34109103
- [Background] Andriessen AE, Eberlein T. Assessment of a wound cleansing solution in the treatment of problem wounds. Wounds. 2008 Jun;20(6):171-5. PMID 25942522
- [Background] Goztok M, Terzi MC, Egeli T, Arslan NC, Canda AE. Does Wound Irrigation with Clorhexidine Gluconate Reduce the Surgical Site Infection Rate in Closure of Temporary Loop Ileostomy? A Prospective Clinical Study. Surg Infect (Larchmt). 2018 Aug/Sep;19(6):634-639. doi: 10.1089/sur.2018.061. Epub 2018 Jul 24. PMID 30040537
- [Background] Chang Z, Liu L, She C, Ren W, Chen H, Zhou C. A meta-analysis examined the effect of stoma on surgical site wound infection in colorectal cancer. Int Wound J. 2023 May;20(5):1578-1583. doi: 10.1111/iwj.14013. Epub 2022 Nov 19. PMID 36401595
- [Background] Nyandoro MG, Seow YT, Stein J, Theophilus M. Single-centre experience of loop ileostomy closure: a retrospective comparison of conventional-linear closure and purse-string closure on surgical-site-infection rates. ANZ J Surg. 2023 Mar;93(3):629-635. doi: 10.1111/ans.18083. Epub 2022 Oct 5. PMID 36197316
- [Background] Zhu Y, Chen J, Lin S, Xu D. Risk factor for the development of surgical site infection following ileostomy reversal: a single-center report. Updates Surg. 2022 Oct;74(5):1675-1682. doi: 10.1007/s13304-022-01335-0. Epub 2022 Aug 24. PMID 36002762
- [Background] Turner MC, Migaly J. Surgical Site Infection: The Clinical and Economic Impact. Clin Colon Rectal Surg. 2019 May;32(3):157-165. doi: 10.1055/s-0038-1677002. Epub 2019 Apr 2. PMID 31061644
- [Background] Wada Y, Miyoshi N, Ohue M, Noura S, Fujino S, Sugimura K, Akita H, Motoori M, Gotoh K, Takahashi H, Kobayashi S, Ohmori T, Fujiwara Y, Yano M. Comparison of surgical techniques for stoma closure: A retrospective study of purse-string skin closure versus conventional skin closure following ileostomy and colostomy reversal. Mol Clin Oncol. 2015 May;3(3):619-622. doi: 10.3892/mco.2015.505. Epub 2015 Feb 6. PMID 26137277
- [Background] Yoon SI, Bae SM, Namgung H, Park DG. Clinical trial on the incidence of wound infection and patient satisfaction after stoma closure: comparison of two skin closure techniques. Ann Coloproctol. 2015 Feb;31(1):29-33. doi: 10.3393/ac.2015.31.1.29. Epub 2015 Feb 28. PMID 25745624
- See also: Related Info — http://creativecommons.org/licenses/by-nc-nd/4.0/